CLINICAL TRIAL: NCT06781307
Title: Department of Nurse-Midwifery and Women Health Graduate Institute of Nurse-Nurse-Midwifery
Brief Title: Effects of Mother-infant Skin-to-skin Contact in Postpartum Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jen-Ai Hospital Institutional Review Board (Industry)
Responsible Party: Principal Investigator, Ming-Chih Chang, Jen-Ai Hospital Principal Investigator, Jen-Ai Hospital Institutional Review Board
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: JenAiH
Record Dates: First submitted 2024-04-06; First posted 2025-01-17 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Attachment
Keywords: Sleep quality; maternal confidence; bonding
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SKIN TO SKIN (Experimental): Daily skin-to skin contact within 30 days of postpartum
  Interventions: Other: skin to skin
- usual care (No Intervention): usual care

INTERVENTIONS:
Other: skin to skin — Intervention measures include 1 hour of skin-to-skin contact between mother and baby every day from day 1 to day 30 postpartum.
  Arms: SKIN TO SKIN

SUMMARY:
When a newborn is delivered in good physiological condition, immediate skin-to-skin contact with the mother is required. Skin-to-skin contact has a wide range of benefits for both mother and baby. The implementation time can start from the birth of the newborn and continue until thereafter. There are benefits both in the short and long term, such as physiological stability, parent-child relationship development, and stability of children's behavioral development. There were 108 cases admitted and the attrition rate was 10%. Therefore, the total number of cases admitted was 118, divided into experimental groups and control groups, and intervention measures were implemented in the experimental group. From the 1st to the 30th day after delivery, there is 1 hour of skin-to-skin contact between mother and baby every day. Fill out the Sleep Quality Visual Analog Scale, Maternal Confidence Scale, and Mother-Infant Bonding Scale on the day after delivery and at one month later.

DETAILED DESCRIPTION:
According to the World Health Organization's clinical care guidelines for childbirth, neonatal care in the third stage of labor: When the newborn is delivered in good physiological condition, it needs to have skin-to-skin contact with the mother immediately. Skin-to-skin contact has extensive benefits for both mother and baby. The implementation time can start from the birth of the newborn and continue thereafter. It has benefits in both the short and long term, such as physiological stability, parent-child relationship development, and child behavioral development stability, etc. Therefore, this study was designed as a quasi-experimental study, using a random method to accept cases. The number of admitted cases was 128, and the attrition rate was 10%. Therefore, the total number of admitted cases was 140, divided into experimental groups and control groups, with intervention measures for the experimental group, and intervention measures. From the 1st to 30th day after delivery, there was 1 hour of skin-to-skin contact between mother and baby every day. On the postpartum day and at the full moon, the sleep quality visual analog scale, maternal confidence scale, and mother-infant bonding scale were filled in, and the statistical method was chi-square. Test, independent sample t test, sample t test, Pearson correlation test, simple regression analysis of the relationship between independent variables and dependent variables and the difference between the experimental group and the control group.

ELIGIBILITY:
Inclusion Criteria:

1. Vaginal delivery to primiparous women
2. Full-term delivery over 37 weeks
3. The pregnancy and delivery process are low-risk cases
4. Can listen, listen, read and write Chinese
5. Agree to participate in this study
6. No mental condition
7. The newborn's vital signs are stable after birth
8. The body appearance is normal after birth and there are no other complications.
9. Can be discharged from hospital together with mother

Exclusion Criteria:

(1)Transfer of newborn to sick nursery after birth

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 70 (Actual)
Dates: Start 2023-11-24 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
sleep quity Visual Analogue Scale | postpartum 30 DAY
  A score of 0 is the worst sleep quality A score Score 10 points for best sleep quality
maternal confidence scale | postpartum 30 DAY
  A score of 0 means never A score of 1 means very little A score of 2 means sometimes A score of 3 mean often A score of 4 mean always The higher the score, the higher the confidence in parenting.
bonding scale | postpartum 30 DAY
  A score of 1 represents strongly disagree, A score of 2 means disagreement, A score of 3 means somewhat disagreeing, A score of 4 means somewhat agree, A score of 5 means agreement A score of 6 means strongly agree The higher the score, the closer the emotional connection between mother and baby.

CONTACTS AND LOCATIONS:
Overall Officials: TSAN-WEN HUANG, college, Study Director — Jen-Ai Hospital Institutional Review Board
Locations (1):
- Jung Ti, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] World Health Organization/UNICEF.(2018). Monitoring the situation of children and Women:Breastfeeding.
- [Background] WHO recommendations on maternal and newborn care for a positive postnatal experience [Internet]. Geneva: World Health Organization; 2022. Available from http://www.ncbi.nlm.nih.gov/books/NBK579657/ PMID 35467813
- [Background] UNICEF(2022) /Too few children benefit from recommended breastfeeding practices
- [Result] Afolabi O, Bunce L, Lusher J, Banbury S. Postnatal depression, maternal-infant bonding and social support: a cross-cultural comparison of Nigerian and British mothers. J Ment Health. 2020 Aug;29(4):424-430. doi: 10.1080/09638237.2017.1340595. Epub 2017 Jul 4. PMID 28675061
- [Result] Aghdas K, Talat K, Sepideh B. Effect of immediate and continuous mother-infant skin-to-skin contact on breastfeeding self-efficacy of primiparous women: a randomised control trial. Women Birth. 2014 Mar;27(1):37-40. doi: 10.1016/j.wombi.2013.09.004. Epub 2013 Nov 9. PMID 24216342
- [Result] Altemus M, Deuster PA, Galliven E, Carter CS, Gold PW. Suppression of hypothalmic-pituitary-adrenal axis responses to stress in lactating women. J Clin Endocrinol Metab. 1995 Oct;80(10):2954-9. doi: 10.1210/jcem.80.10.7559880.
- [Result] Almutairi WM. Literature Review: Physiological Management for Preventing Postpartum Hemorrhage. Healthcare (Basel). 2021 May 31;9(6):658. doi: 10.3390/healthcare9060658. PMID 34073073
- [Result] Badr LK. Further psychometric testing and use of the Maternal Confidence Questionnaire. Issues Compr Pediatr Nurs. 2005 Jul-Sep;28(3):163-74. doi: 10.1080/01460860500227572. PMID 16251162
- [Result] Balatero JS, Spilker AF, McNiesh SG. Barriers to Skin-to-Skin Contact after Cesarean Birth. MCN Am J Matern Child Nurs. 2019 May/Jun;44(3):137-143. doi: 10.1097/NMC.0000000000000521. PMID 31033584
- [Result] Beato AF, Albuquerque S, Komurcu Akik B, da Costa LP, Salvador A. Do Maternal Self-Criticism and Symptoms of Postpartum Depression and Anxiety Mediate the Effect of History of Depression and Anxiety Symptoms on Mother-Infant Bonding? Parallel-Serial Mediation Models. Front Psychol. 2022 May 26;13:858356. doi: 10.3389/fpsyg.2022.858356. eCollection 2022. PMID 35693484
- [Result] Bicking Kinsey C, Hupcey JE. State of the science of maternal-infant bonding: a principle-based concept analysis. Midwifery. 2013 Dec;29(12):1314-20. doi: 10.1016/j.midw.2012.12.019. Epub 2013 Feb 27. PMID 23452661
- [Result] Bieleninik L, Lutkiewicz K, Cieslak M, Preis-Orlikowska J, Bidzan M. Associations of Maternal-Infant Bonding with Maternal Mental Health, Infant's Characteristics and Socio-Demographical Variables in the Early Postpartum Period: A Cross-Sectional Study. Int J Environ Res Public Health. 2021 Aug 12;18(16):8517. doi: 10.3390/ijerph18168517. PMID 34444265
- [Result] Boonstra TW, Stins JF, Daffertshofer A, Beek PJ. Effects of sleep deprivation on neural functioning: an integrative review. Cell Mol Life Sci. 2007 Apr;64(7-8):934-46. doi: 10.1007/s00018-007-6457-8. PMID 17347797
- [Result] Brimdyr K, Stevens J, Svensson K, Blair A, Turner-Maffei C, Grady J, Bastarache L, Al Alfy A, Crenshaw JT, Giugliani ERJ, Ewald U, Haider R, Jonas W, Kagawa M, Lillieskold S, Maastrup R, Sinclair R, Swift E, Takahashi Y, Cadwell K. Skin-to-skin contact after birth: Developing a research and practice guideline. Acta Paediatr. 2023 Aug;112(8):1633-1643. doi: 10.1111/apa.16842. Epub 2023 May 24. PMID 37166443
- [Result] Bystrova K, Matthiesen AS, Vorontsov I, Widstrom AM, Ransjo-Arvidson AB, Uvnas-Moberg K. Maternal axillar and breast temperature after giving birth: effects of delivery ward practices and relation to infant temperature. Birth. 2007 Dec;34(4):291-300. doi: 10.1111/j.1523-536X.2007.00187.x. PMID 18021144
- [Result] Charpak N, de Calume ZF, Ruiz JG. "The Bogota Declaration on Kangaroo Mother Care": conclusions at the second international workshop on the method. Second International Workshop of Kangaroo Mother Care. Acta Paediatr. 2000 Sep;89(9):1137-40. doi: 10.1080/713794578. No abstract available. PMID 11071099
- [Result] Cong S, Wang R, Fan X, Song X, Sha L, Zhu Z, Zhou H, Liu Y, Zhang A. Skin-to-skin contact to improve premature mothers' anxiety and stress state: A meta-analysis. Matern Child Nutr. 2021 Oct;17(4):e13245. doi: 10.1111/mcn.13245. Epub 2021 Jul 13. PMID 34258864
- [Result] Csaszar-Nagy N, Bokkon I. Mother-newborn separation at birth in hospitals: A possible risk for neurodevelopmental disorders? Neurosci Biobehav Rev. 2018 Jan;84:337-351. doi: 10.1016/j.neubiorev.2017.08.013. Epub 2017 Aug 26. PMID 28851575
- [Result] Cuerva MJ, Carbonell M, Boria F, Gil MM, De La Calle M, Bartha JL. Influence on operative time of immediate skin-to-skin care in low-risk primary cesarean births for breech presentation: Retrospective cohort study. Birth. 2023 Sep;50(3):571-577. doi: 10.1111/birt.12683. Epub 2022 Oct 20. PMID 36265127
- [Result] Doyle FL, Dickson SJ, Eapen V, Frick PJ, Kimonis ER, Hawes DJ, Moul C, Richmond JL, Mehta D, Dadds MR. Towards Preventative Psychiatry: Concurrent and Longitudinal Predictors of Postnatal Maternal-Infant Bonding. Child Psychiatry Hum Dev. 2023 Dec;54(6):1723-1736. doi: 10.1007/s10578-022-01365-0. Epub 2022 May 26. PMID 35616764
- [Result] Emmanuel E, Creedy DK, St John W, Gamble J, Brown C. Maternal role development following childbirth among Australian women. J Adv Nurs. 2008 Oct;64(1):18-26. doi: 10.1111/j.1365-2648.2008.04757.x. PMID 18808589
- [Result] El Sehmawy AA, Younes Abd Elaziz S, Elwahed RMA, Elsheikh AA. Skin-to-skin contact and its effect on mothers' postpartum psychological distress and their full-term neonate in Egypt. J Trop Pediatr. 2023 Apr 5;69(3):fmad020. doi: 10.1093/tropej/fmad020. PMID 37203231
- [Result] Feldman R, Magori-Cohen R, Galili G, Singer M, Louzoun Y. Mother and infant coordinate heart rhythms through episodes of interaction synchrony. Infant Behav Dev. 2011 Dec;34(4):569-77. doi: 10.1016/j.infbeh.2011.06.008. Epub 2011 Jul 20. PMID 21767879
- [Result] Friedman M, Hamilton C, Samuelson CG, Kelley K, Taylor D, Pearson-Chauhan K, Maley A, Taylor R, Venkatesan TK. Transoral robotic glossectomy for the treatment of obstructive sleep apnea-hypopnea syndrome. Otolaryngol Head Neck Surg. 2012 May;146(5):854-62. doi: 10.1177/0194599811434262. Epub 2012 Jan 13. PMID 22247514
- [Result] Gray L, Watt L, Blass EM. Skin-to-skin contact is analgesic in healthy newborns. Pediatrics. 2000 Jan;105(1):e14. doi: 10.1542/peds.105.1.e14. PMID 10617751
- [Result] Hairston IS, Handelzalts JE, Lehman-Inbar T, Kovo M. Mother-infant bonding is not associated with feeding type: a community study sample. BMC Pregnancy Childbirth. 2019 Apr 11;19(1):125. doi: 10.1186/s12884-019-2264-0. PMID 30975095
- [Result] Hakanen H, Flykt M, Sinerva E, Nolvi S, Kataja EL, Pelto J, Karlsson H, Karlsson L, Korja R. How maternal pre- and postnatal symptoms of depression and anxiety affect early mother-infant interaction? J Affect Disord. 2019 Oct 1;257:83-90. doi: 10.1016/j.jad.2019.06.048. Epub 2019 Jul 2. PMID 31299408
- [Result] Hall D, Kirsten G. Kangaroo Mother Care--a review. Transfus Med. 2008 Apr;18(2):77-82. doi: 10.1111/j.1365-3148.2007.00812.x. PMID 18399840
- [Result] Hung HM, Chen CH. Sleep quality in postpartum women: exploring correlation with childbirth experience and household work. J Nurs Res. 2014 Mar;22(1):20-7. doi: 10.1097/jnr.0000000000000015. PMID 24517896
- [Result] JayaSalengia B, Rajeswari S, Nalini S. The Relationship between Maternal Confidence, Infant Temperament, and Postpartum Depression. Iran J Nurs Midwifery Res. 2019 Nov 7;24(6):437-443. doi: 10.4103/ijnmr.IJNMR_208_18. eCollection 2019 Nov-Dec. PMID 31772918
- [Result] Karimi FZ, Heidarian Miri H, Salehian M, Khadivzadeh T, Bakhshi M. The Effect of Mother-Infant Skin to Skin Contact after Birth on Third Stage of Labor: A Systematic Review and Meta-Analysis. Iran J Public Health. 2019 Apr;48(4):612-620. PMID 31110971
- [Result] Aydin Kartal Y, Kaya L, Yazici S, Engin B, Karakus R. Effects of skin-to-skin contact on afterpain and postpartum hemorrhage: A randomized controlled trial. Nurs Health Sci. 2022 Jun;24(2):479-486. doi: 10.1111/nhs.12945. Epub 2022 May 9. PMID 35451239
- [Result] Kostandy RR, Ludington-Hoe SM. The evolution of the science of kangaroo (mother) care (skin-to-skin contact). Birth Defects Res. 2019 Sep 1;111(15):1032-1043. doi: 10.1002/bdr2.1565. Epub 2019 Aug 16. PMID 31419082
- [Result] Korukcu O. Psycho-adaptive changes and psychological growth after childbirth in primiparous women. Perspect Psychiatr Care. 2020 Jan;56(1):213-221. doi: 10.1111/ppc.12413. Epub 2019 Jun 21. PMID 31225903
- [Result] Yilmaz Kurt F, Kucukoglu S, Aytekin Ozdemir A, Ogul T, Turkon H, Atay S, Aski N. The effect of kangaroo care on cortisol levels and immune factors in breast milk. Dev Psychobiol. 2023 Jul;65(5):e22402. doi: 10.1002/dev.22402. PMID 37338250
- [Result] Le Bas GA, Youssef GJ, Macdonald JA, Mattick R, Teague SJ, Honan I, McIntosh JE, Khor S, Rossen L, Elliott EJ, Allsop S, Burns L, Olsson CA, Hutchinson DM. Maternal bonding, negative affect, and infant social-emotional development: A prospective cohort study. J Affect Disord. 2021 Feb 15;281:926-934. doi: 10.1016/j.jad.2020.11.031. Epub 2020 Nov 11. PMID 33229017
- [Result] Liu CC, Chen YC, Yeh YP, Hsieh YS. Effects of maternal confidence and competence on maternal parenting stress in newborn care. J Adv Nurs. 2012 Apr;68(4):908-18. doi: 10.1111/j.1365-2648.2011.05796.x. Epub 2011 Jul 27. PMID 21790741
- [Result] Lillieskold S, Zwedberg S, Linner A, Jonas W. Parents' Experiences of Immediate Skin-to-Skin Contact After the Birth of Their Very Preterm Neonates. J Obstet Gynecol Neonatal Nurs. 2022 Jan;51(1):53-64. doi: 10.1016/j.jogn.2021.10.002. Epub 2021 Nov 9. PMID 34767779
- [Result] Linner A, Lode Kolz K, Klemming S, Bergman N, Lillieskold S, Markhus Pike H, Westrup B, Rettedal S, Jonas W. Immediate skin-to-skin contact may have beneficial effects on the cardiorespiratory stabilisation in very preterm infants. Acta Paediatr. 2022 Aug;111(8):1507-1514. doi: 10.1111/apa.16371. Epub 2022 Apr 28. PMID 35466432
- [Result] Maehara K, Mori E, Tsuchiya M, Iwata H, Sakajo A, Tamakoshi K. Factors affecting maternal confidence and satisfaction in older Japanese primiparae during postpartum hospital stay. Int J Nurs Pract. 2016 Apr;22 Suppl 1:14-21. doi: 10.1111/ijn.12435. PMID 27184698
- [Result] Matthiesen AS, Ransjo-Arvidson AB, Nissen E, Uvnas-Moberg K. Postpartum maternal oxytocin release by newborns: effects of infant hand massage and sucking. Birth. 2001 Mar;28(1):13-9. doi: 10.1046/j.1523-536x.2001.00013.x. PMID 11264623
- [Result] McVeigh C. Motherhood experiences from the perspective of first-time mothers. Clin Nurs Res. 1997 Nov;6(4):335-48. doi: 10.1177/105477389700600404. PMID 9384054
- [Result] Medic G, Wille M, Hemels ME. Short- and long-term health consequences of sleep disruption. Nat Sci Sleep. 2017 May 19;9:151-161. doi: 10.2147/NSS.S134864. eCollection 2017. PMID 28579842
- [Result] Mercer RT. Becoming a mother versus maternal role attainment. J Nurs Scholarsh. 2004;36(3):226-32. doi: 10.1111/j.1547-5069.2004.04042.x. PMID 15495491
- [Result] Moberg KU, Handlin L, Petersson M. Neuroendocrine mechanisms involved in the physiological effects caused by skin-to-skin contact - With a particular focus on the oxytocinergic system. Infant Behav Dev. 2020 Nov;61:101482. doi: 10.1016/j.infbeh.2020.101482. Epub 2020 Sep 10. PMID 32919112
- [Result] Nath S, Pearson RM, Moran P, Pawlby S, Molyneaux E, Challacombe FL, Howard LM. The association between prenatal maternal anxiety disorders and postpartum perceived and observed mother-infant relationship quality. J Anxiety Disord. 2019 Dec;68:102148. doi: 10.1016/j.janxdis.2019.102148. Epub 2019 Sep 21. PMID 31604204
- [Result] Ngai FW, Wai-Chi Chan S, Ip WY. Predictors and correlates of maternal role competence and satisfaction. Nurs Res. 2010 May-Jun;59(3):185-93. doi: 10.1097/NNR.0b013e3181dbb9ee. PMID 20404775
- [Result] Nissen E, Lilja G, Widstrom AM, Uvnas-Moberg K. Elevation of oxytocin levels early post partum in women. Acta Obstet Gynecol Scand. 1995 Aug;74(7):530-3. doi: 10.3109/00016349509024384. PMID 7618451
- [Result] Nagasawa M, Okabe S, Mogi K, Kikusui T. Oxytocin and mutual communication in mother-infant bonding. Front Hum Neurosci. 2012 Feb 28;6:31. doi: 10.3389/fnhum.2012.00031. eCollection 2012 Jan 30. PMID 22375116
- [Result] Ngai FW, Chan SW, Holroyd E. Chinese primiparous women's experiences of early motherhood: factors affecting maternal role competence. J Clin Nurs. 2011 May;20(9-10):1481-9. doi: 10.1111/j.1365-2702.2010.03415.x. Epub 2011 Feb 8. PMID 21299660
- [Result] Nolvi S, Karlsson L, Bridgett DJ, Pajulo M, Tolvanen M, Karlsson H. Maternal postnatal psychiatric symptoms and infant temperament affect early mother-infant bonding. Infant Behav Dev. 2016 May;43:13-23. doi: 10.1016/j.infbeh.2016.03.003. Epub 2016 Apr 4. PMID 27054496
- [Result] O'Dea GA, Youssef GJ, Hagg LJ, Francis LM, Spry EA, Rossen L, Smith I, Teague SJ, Mansour K, Booth A, Davies S, Hutchinson D, Macdonald JA. Associations between maternal psychological distress and mother-infant bonding: a systematic review and meta-analysis. Arch Womens Ment Health. 2023 Aug;26(4):441-452. doi: 10.1007/s00737-023-01332-1. Epub 2023 Jun 15. PMID 37316760
- [Result] Ohara M, Okada T, Kubota C, Nakamura Y, Shiino T, Aleksic B, Morikawa M, Yamauchi A, Uno Y, Murase S, Goto S, Kanai A, Masuda T, Ando M, Ozaki N. Relationship between maternal depression and bonding failure: A prospective cohort study of pregnant women. Psychiatry Clin Neurosci. 2017 Oct;71(10):733-741. doi: 10.1111/pcn.12541. Epub 2017 Jul 7. PMID 28556440
- [Result] Owais S, Chow CHT, Furtado M, Frey BN, Van Lieshout RJ. Non-pharmacological interventions for improving postpartum maternal sleep: A systematic review and meta-analysis. Sleep Med Rev. 2018 Oct;41:87-100. doi: 10.1016/j.smrv.2018.01.005. Epub 2018 Jan 31. PMID 29449122
- [Result] Owusu-Ansah FE, Bigelow AE, Power M. The effect of mother-infant skin-to-skin contact on Ghanaian infants' response to the Still Face Task: Comparison between Ghanaian and Canadian mother-infant dyads. Infant Behav Dev. 2019 Nov;57:101367. doi: 10.1016/j.infbeh.2019.101367. Epub 2019 Oct 23. PMID 31654883
- [Result] Pang KP, Terris DJ. Modified cautery-assisted palatal stiffening operation: new method for treating snoring and mild obstructive sleep apnea. Otolaryngol Head Neck Surg. 2007 May;136(5):823-6. doi: 10.1016/j.otohns.2006.11.014. PMID 17478223
- [Result] Pados BF, Hess F. Systematic Review of the Effects of Skin-to-Skin Care on Short-Term Physiologic Stress Outcomes in Preterm Infants in the Neonatal Intensive Care Unit. Adv Neonatal Care. 2020 Feb;20(1):48-58. doi: 10.1097/ANC.0000000000000596. PMID 30893092
- [Result] Rafii F, Alinejad-Naeini M, Peyrovi H. Maternal Role Attainment in Mothers with Term Neonate: A Hybrid Concept Analysis. Iran J Nurs Midwifery Res. 2020 Jun 17;25(4):304-313. doi: 10.4103/ijnmr.IJNMR_201_19. eCollection 2020 Jul-Aug. PMID 33014742
- [Result] Ruiz MT, Azevedo NF, Raponi MBG, Fonseca LMM, Wernet M, Silva MPC, Contim D. Skin-to-Skin Contact in the Third Stage of Labor and Postpartum Hemorrhage Prevention: A Scoping Review. Matern Child Health J. 2023 Apr;27(4):582-596. doi: 10.1007/s10995-022-03582-4. Epub 2023 Mar 3. PMID 36867304
- [Result] Saxton A, Fahy K, Rolfe M, Skinner V, Hastie C. Does skin-to-skin contact and breast feeding at birth affect the rate of primary postpartum haemorrhage: Results of a cohort study. Midwifery. 2015 Nov;31(11):1110-7. doi: 10.1016/j.midw.2015.07.008. Epub 2015 Jul 29. PMID 26277824
- [Result] Sehgal A, Nitzan I, Jayawickreme N, Menahem S. Impact of Skin-to-Skin Parent-Infant Care on Preterm Circulatory Physiology. J Pediatr. 2020 Jul;222:91-97.e2. doi: 10.1016/j.jpeds.2020.03.041. Epub 2020 May 7. PMID 32389414
- [Result] Shreffler KM, Spierling TN, Jespersen JE, Tiemeyer S. Pregnancy intendedness, maternal-fetal bonding, and postnatal maternal-infant bonding. Infant Ment Health J. 2021 May;42(3):362-373. doi: 10.1002/imhj.21919. Epub 2021 Apr 15. PMID 33860552
- [Result] Stevens J, Schmied V, Burns E, Dahlen HG. Skin-to-skin contact and what women want in the first hours after a caesarean section. Midwifery. 2019 Jul;74:140-146. doi: 10.1016/j.midw.2019.03.020. Epub 2019 Mar 27. PMID 30954633
- [Result] Stevens J, Schmied V, Burns E, Dahlen HG. Who owns the baby? A video ethnography of skin-to-skin contact after a caesarean section. Women Birth. 2018 Dec;31(6):453-462. doi: 10.1016/j.wombi.2018.02.005. Epub 2018 Mar 2. PMID 29496385
- [Result] Tognasso G, Gorla L, Ambrosini C, Figurella F, De Carli P, Parolin L, Sarracino D, Santona A. Parenting Stress, Maternal Self-Efficacy and Confidence in Caretaking in a Sample of Mothers with Newborns (0-1 Month). Int J Environ Res Public Health. 2022 Aug 5;19(15):9651. doi: 10.3390/ijerph19159651. PMID 35955005
- [Result] Uvnas-Moberg K. Neuroendocrinology of the mother-child interaction. Trends Endocrinol Metab. 1996 May-Jun;7(4):126-31. doi: 10.1016/1043-2760(96)00036-7. PMID 18406738
- [Result] Vargas-Porras C, Roa-Diaz ZM, Hernandez-Hincapie HG, Ferre-Grau C, de Molina-Fernandez MI. Efficacy of a multimodal nursing intervention strategy in the process of becoming a mother: A randomized controlled trial. Res Nurs Health. 2021 Jun;44(3):424-437. doi: 10.1002/nur.22123. Epub 2021 Mar 8. PMID 33682146
- [Result] Vecsey CG, Baillie GS, Jaganath D, Havekes R, Daniels A, Wimmer M, Huang T, Brown KM, Li XY, Descalzi G, Kim SS, Chen T, Shang YZ, Zhuo M, Houslay MD, Abel T. Sleep deprivation impairs cAMP signalling in the hippocampus. Nature. 2009 Oct 22;461(7267):1122-5. doi: 10.1038/nature08488. PMID 19847264
- [Result] Vittner D, McGrath J, Robinson J, Lawhon G, Cusson R, Eisenfeld L, Walsh S, Young E, Cong X. Increase in Oxytocin From Skin-to-Skin Contact Enhances Development of Parent-Infant Relationship. Biol Res Nurs. 2018 Jan;20(1):54-62. doi: 10.1177/1099800417735633. Epub 2017 Oct 11. PMID 29017336
- [Result] Vittner D, Butler S, Smith K, Makris N, Brownell E, Samra H, McGrath J. Parent Engagement Correlates With Parent and Preterm Infant Oxytocin Release During Skin-to-Skin Contact. Adv Neonatal Care. 2019 Feb;19(1):73-79. doi: 10.1097/ANC.0000000000000558. PMID 30335622
- [Result] Winberg J. Mother and newborn baby: mutual regulation of physiology and behavior--a selective review. Dev Psychobiol. 2005 Nov;47(3):217-29. doi: 10.1002/dev.20094. PMID 16252290
- [Result] Widstrom AM, Lilja G, Aaltomaa-Michalias P, Dahllof A, Lintula M, Nissen E. Newborn behaviour to locate the breast when skin-to-skin: a possible method for enabling early self-regulation. Acta Paediatr. 2011 Jan;100(1):79-85. doi: 10.1111/j.1651-2227.2010.01983.x. Epub 2010 Sep 14. PMID 20712833
- [Result] Widstrom AM, Brimdyr K, Svensson K, Cadwell K, Nissen E. Skin-to-skin contact the first hour after birth, underlying implications and clinical practice. Acta Paediatr. 2019 Jul;108(7):1192-1204. doi: 10.1111/apa.14754. Epub 2019 Mar 13. PMID 30762247
- [Result] Weisman O, Zagoory-Sharon O, Feldman R. Oxytocin administration to parent enhances infant physiological and behavioral readiness for social engagement. Biol Psychiatry. 2012 Dec 15;72(12):982-9. doi: 10.1016/j.biopsych.2012.06.011. Epub 2012 Jul 13. PMID 22795645
- [Result] World Health Organization.(2022). WHO advises immediate skin to skin care for survival of small and preterm babies.

DOCUMENTS (1):
  • Informed Consent Form (2023-11-25): https://cdn.clinicaltrials.gov/large-docs/07/NCT06781307/ICF_000.pdf